CLINICAL TRIAL: NCT01173471
Title: A Double Masked, Placebo Controlled, Randomised, Parallel Group Phase IIa Study to Assess the Tolerability, Safety, and Efficacy of AZD4017 for Raised Intra-Ocular Pressure
Brief Title: A Phase IIa Study to Assess the Tolerability, Safety, and Efficacy of AZD4017 for Raised Intra-ocular Pressure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D4250C00001; 2010-020932-20 (EudraCT Number)
Record Dates: First submitted 2010-07-29; First posted 2010-08-02 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-01

CONDITIONS: Raised Intraocular Pressure
Keywords: Raised intraocular pressure
MeSH Terms: conditions — Ocular Hypertension | interventions — 2-(1-(5-(cyclohexylcarbamoyl)-6-propylsulfanylpyridin-2-yl)-3-piperidyl)acetic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1) AZD4017 (Experimental): Europe: 200 mg AZD4017
  Interventions: Drug: AZD4017
- 2) Placebo (Placebo Comparator): Europe: placebo
  Interventions: Drug: Placebo
- 3) AZD4017 (Experimental): USA: 800 mg AZD4017
  Interventions: Drug: AZD4017
- 4) Placebo (Placebo Comparator): USA: placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD4017 — tablet, oral, one tablet once daily, 28 days
  Arms: 1) AZD4017
Drug: Placebo — matching placebo tablet, oral, one tablet once daily, 28 days
  Arms: 2) Placebo
Drug: AZD4017 — tablet, oral 2 tablets twice daily, 28 days
  Arms: 3) AZD4017
Drug: Placebo — matching placebo tablets, oral, 2 tablets twice daily, 28 days
  Arms: 4) Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of systemically administered AZD4017, compared with placebo, over a 28-day period in patients with raised intra-ocular pressure (IOP).

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of intra-ocular hypertension (raised IOP), or primary open-angle glaucoma (POAG), with IOP >20 mmHg and ≤36 mmHg in the study eye, and is currently prescribed a stable dose of a single anti-glaucoma medication that began at least 30 days prior to the screening visit; OR
* Must have a diagnosis of intra-ocular hypertension (raised IOP), defined as an IOP ≥22 mmHg and ≤36 mmHg in the study eye while not on anti-glaucoma medication
* Male patients must be willing to use barrier contraception with spermicide, ie, condoms, from the day of first dosing until 3 months after dosing with IP
* Placebo treatment for duration of the study must not be considered detrimental to the patient

Exclusion Criteria:

* Have uncontrolled intra-ocular hypertension (>36 mmHg)
* Have experienced a significant visual field loss or showed evidence of progressive visual field loss within the last year (as defined by >1 dB/yr average loss or vision threatening new defect)
* Have had severe eye trauma at any time

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Bryson, PhD, Study Director — AstraZeneca R&D; Tony Ho, MD, Study Director — AstraZeneca R&D
Locations (11):
- United States (7):
  - Research Site, Newport Beach, California
  - Research Site, Atlanta, Georgia
  - Research Site, Morrow, Georgia
  - Research Site, Overland Park, Kansas
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Memphis, Tennessee
- Sweden (3):
  - Research Site, Lund
  - Research Site, Mölndal
  - Research Site, Stockholm
- Research Site, Nottingham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted in 19 centers in the US, UK, and Sweden between 13 December 2010 and 06 November 2012. A total of 117 patients were screened in the study and of these, 50 were randomized into the double-blind treatment period.
Pre-assignment Details: Diagnosis of intra-ocular hypertension (raised IOP), or POAG, with IOP >20 mmHg and =<36 mmHg, and currently prescribed a stable dose of one anti-glaucoma medication that began at least 30 days prior to the screening visit or a diagnosis of intra-ocular hypertension, defined as an IOP >22 mmHg and =<36 mmHg while not on anti-glaucoma medication.
Groups:
- Placebo OD: Placebo once daily
- AZD4017 200 mg OD: AZD4017 200 mg once daily
- Placebo BID: Placebo twice daily
- AZD4017 400 mg BID: AZD4017 400 mg twice daily
Period: Overall Study
Arm/Group | Placebo OD | AZD4017 200 mg OD | Placebo BID | AZD4017 400 mg BID
Started | 6 (Randomized) | 7 (Randomized) | 18 (Randomized) | 19 (Randomized)
Received Treatment | 6 | 7 | 18 | 19
Completed Treatment | 4 | 7 | 15 | 18
Completed | 4 (Completed study) | 7 (Completed study) | 15 (Completed study) | 18 (Completed study)
Not Completed | 2 | 0 | 3 | 1
Not completed — Eligibility criteria not fulfilled | 0 | 0 | 1 | 1
Not completed — Condition under investigation worsened | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Reason given as Other | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo OD | AZD4017 200 mg OD | Placebo BID | AZD4017 400 mg BID | Total
Number analyzed (Participants) | 6 | 7 | 18 | 19 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63 (6.7) | 63 (8.7) | 57 (15.1) | 65 (10.1) | 61 (11.9)
Age, Customized [Number; unit: Participants]
  <50 years | 0 | 1 | 5 | 2 | 8
  >=50-<65 years | 3 | 4 | 6 | 5 | 18
  >=65 years | 3 | 2 | 7 | 12 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 9 | 11 | 25
  Male | 4 | 4 | 9 | 8 | 25
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 5 | 5 | 10
  White | 6 | 7 | 12 | 14 | 39
  Other | 0 | 0 | 0 | 0 | 0
  Missing | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United Kingdom | 2 | 4 | 0 | 0 | 6
  Sweden | 4 | 3 | 0 | 0 | 7
  United States | 0 | 0 | 18 | 19 | 37
Stratification factor [Number; unit: Participants]
  Add-on to intra-ocular pressure medication | 0 | 1 | 8 | 9 | 18
  Not on intra-ocular pressure medication | 6 | 6 | 10 | 10 | 32

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Mean Intra-ocular Pressure Compared With Baseline After 4 Weeks Treatment
Time Frame: Baseline to 4 weeks
Population: Efficacy analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo OD | AZD4017 200 mg OD | Placebo BID | AZD4017 400 mg BID
Number analyzed (Participants) | 6 | 7 | 16 | 19
Percentage change | 0.8 [-15.6 to 17.3] | -0.4 [-13.8 to 13.0] | -8.1 [-13.3 to -2.9] | -11.0 [-15.8 to -6.2]
Statistical Analysis 1: Comparison: Placebo OD vs AZD4017 200 mg OD; Test type: Superiority or Other; p = 0.822, Mixed Models Analysis; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-15.2 to 12.6], Standard Error of Mean 5.352 — Difference is (AZD4017 200 mg OD - Placebo OD)
Statistical Analysis 2: Comparison: Placebo BID vs AZD4017 400 mg BID; Test type: Superiority or Other; p = 0.413, Mixed Models Analysis; Mean Difference (Final Values) = -2.9, 95% CI 2-sided [-10.1 to 4.3], Standard Error of Mean 3.516 — Difference is (AZD4017 400 mg BID - Placebo BID)

2. Secondary Outcome: Clinically Relevant Change in Intra-ocular Pressure After 4 Weeks of Treatment
Time Frame: Baseline to 4 weeks
Population: Efficacy analysis set
Measure: Number; unit: Participants
Arm/Group | Placebo OD | AZD4017 200 mg OD | Placebo BID | AZD4017 400 mg BID
Number analyzed (Participants) | 6 | 7 | 18 | 19
Participants
  >= 20% decrease in intra-ocular pressure | 0 | 0 | 1 | 4
  >= 30% decrease in intra-ocular pressure | 0 | 0 | 0 | 0

3. Secondary Outcome: Change in Mean Intra-ocular Pressure Compared With Baseline After 4 Weeks Treatment
Time Frame: Baseline to 4 weeks
Population: Efficacy analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Placebo OD | AZD4017 200 mg OD | Placebo BID | AZD4017 400 mg BID
Number analyzed (Participants) | 6 | 7 | 16 | 19
mmHg | 0.1 [-4.8 to 4.9] | -0.4 [-4.4 to 3.5] | -1.9 [-3.3 to -0.6] | -2.6 [-3.8 to -1.3]
Statistical Analysis 1: Comparison: Placebo OD vs AZD4017 200 mg OD; Test type: Superiority or Other; p = 0.758, Mixed Models Analysis; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-4.8 to 3.7], Standard Error of Mean 1.570 — Difference is (AZD4017 200 mg OD - Placebo OD)
Statistical Analysis 2: Comparison: Placebo BID vs AZD4017 400 mg BID; Test type: Superiority or Other; p = 0.467, Mixed Models Analysis; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-2.5 to 1.2], Standard Error of Mean 0.909 — Difference is (AZD4017 400 mg BID - Placebo BID)

ADVERSE EVENTS:
Time Frame: 4-week treatment period.
Description: All patients were required to return for a mandatory follow-up visit (Visit 8) between 14 and 21 days, inclusive, after the last dose of study medication. Any ongoing adverse events (AEs) at the follow-up visit were followed until resolution, until the AE stabilized, until it was otherwise explained, or until the patient was lost to follow-up.
Arm/Group | Placebo OD | AZD4017 200 mg OD | Placebo BID | AZD4017 400 mg BID
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 5/6 | 3/7 | 5/18 | 7/19
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo OD (N=6) | AZD4017 200 mg OD (N=7) | Placebo BID (N=18) | AZD4017 400 mg BID (N=19)
ASYMPTOMATIC BACTERIURIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONJUNCTIVITIS INFECTIVE (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFECTED BITES (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BALANCE DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLEPHARITIS (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONJUNCTIVAL HYPERAEMIA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DELLEN (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DRY EYE (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EYE PAIN (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PHOTOPHOBIA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VITREOUS DETACHMENT (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FLUSHING (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LIP PRURITUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SENSATION OF HEAVINESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
INTRAOCULAR PRESSURE INCREASED (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
JOINT INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor recognises that the Trust and Investigator have a responsibility under the Research Governance Framework for Health and Social Care to ensure that results of scientific interest arising from the Clinical Trial are appropriately published and disseminated. Such data will be submitted to the Sponsor for review and comment prior to publication. The Trust agrees, and shall ensure that the Investigator agrees, that all reasonable comments made by the Sponsor will be incorporated.